CLINICAL TRIAL: NCT04534738
Title: Diet And Nutrition In CAncer (The DANICA Study): The Effect of a Mediterranean Diet Intervention on Cancer-related Fatigue and Mitochondrial Function During Chemotherapy
Brief Title: The Effect of a Mediterranean Diet Intervention on Cancer-related Fatigue and Mitochondrial Function During Chemotherapy
Acronym: DANICA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS20082
Record Dates: First submitted 2020-08-17; First posted 2020-09-01 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: nutrition; diet
MeSH Terms: conditions — Neoplasms | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): Participants in the Mediterranean Diet arm are asked to follow a Mediterranean Diet for 8 weeks. The diet is ad libitum. A combination of fresh, frozen, and shelf-stable meals are provided for the first 4 weeks. Also during the first 4 weeks, participants receive an education session to discuss how to effectively implement a Mediterranean Diet into their daily routine.
  Interventions: Behavioral: Mediterranean Diet
- Usual care (No Intervention): Participants in the usual care are will complete all the same study assessments as those in the intervention group. They will not receive any specific dietary advice, but they will be permitted to seek dietary advice outside the study. Data from this group are indispensable in understanding the nutritional habits and preferences of patients undergoing chemotherapy, and these data will be used to optimize nutritional interventions in future studies. At the end of the 8-week intervention, the participants in the usual care group will be provided the intervention materials gratis, including one-week of Mediterranean Diet food and education materials.

INTERVENTIONS:
Behavioral: Mediterranean Diet — The Mediterranean Diet is high in fruit, vegetables, legumes, nuts and seeds, whole grains, and olive oil; moderate in seafood, dairy products (e.g., cheese and yogurt but not whole milk or butter), eggs, poultry, and red wine with meals; and low consumption of sweet desserts, red meat, and highly processed foods.
  Arms: Mediterranean Diet

SUMMARY:
This study will assess the feasibility of delivering an 8-week Mediterranean Diet intervention as well as the intervention's preliminary efficacy on cancer-related fatigue among patients undergoing chemotherapy, compared to usual care. In the first 4 weeks of the intervention, we will provide the participants with food and educate them on the principles and components of the Mediterranean Diet, while in the second 4 weeks participants will prepare their own food. In addition, we will evaluate changes in metabolism and mitochondrial function during 4 weeks of chemotherapy and determine how adherence to a Mediterranean diet modulates these changes during these 4 weeks.

The hypothesis is that the intervention will promote adherence to the Mediterranean Diet. The second hypothesis is that adherence will be associated with alleviation of fatigue and improvements in metabolic and mitochondrial function.

ELIGIBILITY:
Inclusion Criteria (Participants must…):

* Have a diagnosis of cancer,
* Be scheduled to receive chemotherapy and have at least 6 weeks remaining,
* Be able to speak English,
* Be willing to adhere to study procedures, and
* Be able to provide written informed consent.

Exclusion Criteria (Participants must not…):

* Be on enteral or parenteral nutrition,
* Be pregnant,
* Have distant metastases,
* Have a brain tumor,
* Have any plan to get radiation to the head,
* Have specific dietary needs that a Mediterranean diet cannot meet (e.g., allergies to nuts, gluten intolerance), or already be following the Mediterranean diet (i.e., have a score ≥10 on a modified 14-item Mediterranean Diet questionnaire).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber S. Kleckner, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Pluta Cancer Center, Rochester, New York
  - Wilmot Cancer Institute, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mediterranean Diet | Usual Care
Started | 23 | 10
Completed | 23 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mediterranean Diet | Usual Care | Total
Number analyzed (Participants) | 23 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.2) | 49.2 (16.3) | 51.0 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 9 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 10 | 33
Type of cancer [Count of Participants; unit: Participants]
  Breast cancer | 20 | 10 | 30
  Other | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Enrolled Completed the Study.
Description: To assess feasibility of the study, we will report what percentage of patients who enrolled completed the study.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mediterranean Diet | Usual Care
Number analyzed (Participants) | 23 | 10
Participants | 23 | 10

2. Primary Outcome: Scores From the 14-item Mediterranean Diet Questionnaire
Description: In order to assess adherence to the diet, we will report scores from the 14-item Mediterranean Diet questionnaire at 8 weeks. Scores range from 0 to 14 points. A higher score indicates greater adherence to the Mediterranean Diet.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mediterranean Diet | Usual Care
Number analyzed (Participants) | 23 | 10
units on a scale | 6.5 (2.6) | 5.2 (3.0)

3. Secondary Outcome: The Functional Assessment of Chronic Illness-Fatigue (FACIT-F) Questionnaire
Description: Fatigue will be measured using the Functional Assessment of Chronic Illness-Fatigue (FACIT-F). This is a 40-item questionnaire in which a higher score indicates greater well-being. Scores range from 0-160.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mediterranean Diet | Usual Care
Number analyzed (Participants) | 23 | 10
units on a scale | 114.1 (28.4) | 116.9 (20.4)

4. Secondary Outcome: The Functional Assessment of Chronic Illness-Fatigue (FACIT-F) Questionnaire, Fatigue Subscale
Description: Fatigue will be measured using the Functional Assessment of Chronic Illness-Fatigue (FACIT-F), fatigue subscale. This is a 13-item subscale of the FACIT-F questionnaire in which a higher score indicates less fatigue. Scores range from 0-52.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mediterranean Diet | Usual Care
Number analyzed (Participants) | 23 | 10
units on a scale | 35.3 (12.1) | 36.0 (9.8)

ADVERSE EVENTS:
Time Frame: 9-week study
Arm/Group | Mediterranean Diet | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/23 | 2/10
Other Adverse Events (participants affected / at risk) | 0/23 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mediterranean Diet (N=23) | Usual Care (N=10)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — not attributed to the intervention, participant continued with study
Fainting (General disorders) | 1 (1) | 0 (0) — occurred after consent but before randomization and therefore before the start of the intervention, participant continued with study
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) — Not attributed to the intervention, participant continued with study
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Not attributed to the intervention, participant continued with study
Dental infection (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not attributed to the intervention, participant continued with study
Neutropenic fever (General disorders) | 1 (1) | 0 (0) — Not attributed to the intervention, participant continued with study
Cellulitis of the chest wall (General disorders) | 1 (1) | 0 (0) — Not attributed to the intervention, participant continued with study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04534738/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04534738/ICF_001.pdf